CLINICAL TRIAL: NCT05109624
Title: Is Prolonged Period of Prone Position Effective and Safe in Mechanically Ventilated Patients With SARS-COV-2? A Randomized Clinical Trial
Brief Title: Is Prolonged Period of Prone Position Effective and Safe in Mechanically Ventilated Patients With SARS-COV-2?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr Fouad, lecturer of anesthesia and intensive care, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R 160 / 2021
Record Dates: First submitted 2021-11-03; First posted 2021-11-05 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group(A) control group (No Intervention): pronation cycles each last for 16 hours every 24 hours
- group(B) (Active Comparator): pronation cycles each last for 24 hours followed by 6 hours supine position
  Interventions: Procedure: prolonged prone position ventilation

INTERVENTIONS:
Procedure: prolonged prone position ventilation — patients mechanically ventilated with SARS COV 2 will be subjected to a longer than usual period of prone position ventilation
  Arms: group(B)

SUMMARY:
the aim of the study is to assess safety and efficacy of prone position ventilation beyond the usual 16 hrs in patients with SARS-COV-2

ELIGIBILITY:
Inclusion Criteria:

* - American Society of Anesthesiologists (ASA) physical status II- III.
* Sex (male and females).
* Age 18 -80 years.
* Sever adult respiratory distress (ARDS) (defined as a PaO2:FiO2 ratio of <150 mm Hg, with a fraction of inspired oxygen (FiO2) of ≥0.6, a positive end expiratory pressure (PEEP) of ≥5 CmH2O, and a tidal volume of 6 ml/Kg of predicted body weight
* mechanical ventilation for less than 36 hours

Exclusion Criteria:

* - Contraindication for prone positioning

  * increased intracranial tension.
  * face trauma or surgery.
  * Recent Deep venous thrombosis
  * Unstable spine, femur, or pelvic fractures
  * Mean arterial pressure < 65 mm Hg
  * Pregnant women
  * Pneumothorax
  * Prone positioning before inclusion
* Those returned to supine position before completing the session time

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
rate of successful weaning | 28 days
  how many patients successfully extubated, hospital survival, ICU stay
Incidence of complications | 28 days
  Incidence of facial edema, pressure wounds, lines disconnections, hemodynamic instability

SECONDARY OUTCOMES:
Efficacy of oxygenation | 28 days
  mean value of change in PaO2/FiO2 ratio and static lung compliance before and after 3 successive proning cycles

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt